CLINICAL TRIAL: NCT03510871
Title: Nivolumab Plus Ipilimumab as Neoadjuvant Therapy for Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); National Cheng-Kung University Hospital (Other); China Medical University Hospital (Other); Chang Gung Memorial Hospital (Other); Mackay Memorial Hospital (Other); Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2217
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: neoadjuvant therapy; immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nivolumab plus ipilimumab (Experimental): nivolumab plus ipilimumab
  Interventions: Drug: nivolumab, ipilimumab

INTERVENTIONS:
Drug: nivolumab, ipilimumab — All enrolled subjects will receive nivolumab 3 mg/kg plus ipilimumab 1 mg/kg intravenously on day 1 of each cycle (every 3 weeks). Tumor assessment will be done after 6 weeks (2 cycles) and 12 weeks (4 cycles).
  Other Names: nivolumab plus ipilimumab

SUMMARY:
Objectives:

1. To evaluate the efficacy, in terms of tumor shrinkage, objective response rate, and down-stage rate, of nivolumab + ipilimumab as neoadjuvant therapy for patients with HCC;
2. To evaluate the safety profile in patients with HCC who receive neoadjuvant nivolumab + ipilimumab treatment;
3. To collect HCC tumor tissue and peripheral blood samples from the patients for a comprehensive biomarker evaluation for nivolumab + ipilimumab immunotherapy.

DETAILED DESCRIPTION:
Immune checkpoint inhibitor therapy represents the major breakthrough of anticancer drug therapy development in recent years. Inhibitors targeting the cytotoxic T-lymphocyte antigen 4 (CTLA-4) or the programmed death-1 (PD-1) checkpoints have shown antitumor activity in multiple cancer types. Combination of anti-CTLA-4 and anti-PD-1 therapy may increase the objective response rate for patients with advanced cancers and thus may further improve the treatment efficacy. The anti-PD-1 drug nivolumab recently got approval by US FDA for the treatment of advanced hepatocellular carcinoma (HCC) patients who have been treated with sorafenib. Preliminary data also suggested that combination of nivolumab and anti-CTLA-4 therapy could increase the objective response rate for advanced HCC, with a better safety profile compared with conventional combination therapies (cytotoxic chemotherapy or molecular targeted therapy). This project aims to explore whether the high response rate produced by the combination of anti-PD-1 and anti-CTLA-4 may improve the treatment efficacy of HCC patients who are potentially eligible for curative surgery.

This is a single-arm, open-label trial. Eligible subjects must have histological diagnosis of HCC and fulfilling one of the following criteria of 'potentially eligible for curative surgery': (a) AJCC T3 tumor(s) (tumor with macrovascular invasion); (b) AJCC T2 tumors with multiple tumors and bilateral lobes involvement, none more than 5 cm; (c) AJCC T2 tumors with tumor number > 3, none more than 5 cm; (d) AJCC T2 tumors with multiple tumors none more than 5 cm, with significant portal hypertension (splenomegaly, esophageal varices or platelet < 100,000/μL); or (e) solitary tumor > 5 cm, with significant portal hypertension (splenomegaly, esophageal varices or platelet < 100,000/μL) ; (f) Other conditions that are considered high-risk for recurrence after surgery, e.g., direct diaphragmic invasion suspected by imaging。Eligible subjects must have ECOG performance status 0 or 1, Child-Pugh class A liver function, and measurable tumors (by RECIST 1.1). All enrolled subjects will receive nivolumab 3 mg/kg plus ipilimumab 1 mg/kg intravenously on day 1 of each cycle (every 3 weeks). Tumor assessment will be done after 6 weeks (2 cycles) and 12 weeks (4 cycles). Subjects who are considered eligible for curative surgery will receive surgery, while those considered not eligible for surgery will receive other anti-cancer therapy according to current practice guidelines (e.g., trans-catheter arterial chemoembolization). Samples will be collected from the subjects' tumor tissue, peripheral blood, and stool for studies of immune biomarkers.

The primary endpoint is the percentage of subjects with tumor shrinkage (> 10% of decrease of the sum of the target lesions according to RECIST 1.1) after study drug treatment. It is estimated that about 30-50% subjects may have tumor shrinkage after 2-4 cycles of nivolumab + ipilimumab treatment. With type 1 error 0.05；power=0.9，P0=0.30, P1=0.55 respectively, 40 evaluable subjects (subjects who receive at least 2 cycles of study drug treatment and receive the first scheduled assessment of tumor response, assuming a 10% dropout rate) will be required. The study is expected to complete enrollment in 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of HCC with potential for curative surgical resection fulfilling one of the following criteria:

   (A)Tumor(s) with macrovascular invasion. (B)Tumors with one of the following features: (B1)multiple tumors and bilateral lobes involvement, none more than 5 cm (B2)tumor number > 3, none more than 5 cm (B3)multiple tumors none more than 5 cm, with significant portal hypertension (splenomegaly, esophageal varices or platelet < 100,000/μL) (B4)solitary tumor > 5 cm, with significant portal hypertension (splenomegaly, esophageal varices or platelet < 100,000/μL) (B5)Other conditions that are considered high-risk for recurrence after surgery, e.g., direct diaphragmic invasion suspected by imaging。
2. No evidence of extra-hepatic metastases.
3. At least one measurable tumor, according to RECIST version 1.1, that has not been treated with any local procedure.
4. Prior percutaneous ethanol injection, radiofrequency ablation, transarterial embolization, or cryotherapy are allowed if aforementioned local therapy is given at least 4 weeks prior to enrollment and progressive or recurrent disease is documented.
5. Age >= 20 years old.
6. ECOG performance status 0 or 1.
7. Child-Pugh class A liver function.
8. WBC >=2,000/uL (stable, off any growth factor within 4 weeks of study drug administration) ; Platelet>= 60,000/uL.
9. Liver transaminases (ALT and AST) <= 5 times upper limit of normal values (ULN); total bilirubin <=1.5 times ULN; serum creatinine<=1.5 times ULN; creatinine clearance > 50 mL/min (calculated by Cockcroft-Gault formula)
10. Subjects with chronic hepatitis B virus infection (HBV surface antigen (HBsAg) positive) must start antiviral therapy with nucleoside analogs (e.g., entecavir or tenofovir, according to current practice guidelines) before start of study drug treatment.
11. Signed informed consent.

Exclusion Criteria:

1. Receiving concurrent anti-cancer therapy for HCC, which includes local therapy, systemic therapy, or other experimental therapy.
2. Local treatment including radiotherapy (except palliative radiotherapy), percutaneous ethanol injection, radiofrequency ablation, or transarterial embolization administered within 4 weeks prior to enrollment.
3. Major surgical procedure within 2 weeks or minor surgical procedure within 1 week prior to enrollment.
4. History of esophageal/gastric varices or active peptic ulcers that are considered to have high risk of bleeding.
5. History of upper gastrointestinal bleeding within 1 year.
6. Known human immunodeficiency virus (HIV) infection.
7. Major systemic diseases that the investigator considers inappropriate for participation.
8. History of other malignancies except those treated with curative intent for skin cancer (other than melanoma), in situ breast or in situ cervical cancer, or those treated with curative intent for any other cancer with no evidence of disease for 2 years.
9. Any active autoimmune disease or history of known autoimmune disease except for vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
10. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
11. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways).
12. Requirement of systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
13. Prior organ allograft or allogeneic bone marrow transplantation.
14. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
the percentage of subjects with tumor shrinkage after study drug treatment | 4 years
  > 10% of decrease of the sum of the target lesions according to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Wu Liu, MD, PhD, Study Chair — Taiwan Cooperative Oncology Group, NHRI; Chiun Hsu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (8):
- Taiwan (8):
  - Chang-Gung Memorial Hospital, Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang-Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No
Invetigator Initial Trial

REFERENCES:
- [Derived] Lin YJ, Ou DL, Su YY, Hsu CL, Hsiao CF, Ko BS, Chen SC, Wang HW, Wang JH, Wu YM, Jeng YM, Lee WC, Chou SC, Chen TW, Chiu CF, Lin JS, Hsieh CH, Lee CC, Shan YS, Cheng AL, Chen LT, Hsu C. Nivolumab plus ipilimumab for potentially resectable hepatocellular carcinoma: Long-term efficacy and biomarker exploration. J Hepatol. 2026 Feb;84(2):316-328. doi: 10.1016/j.jhep.2025.08.035. Epub 2025 Sep 17. PMID 40972843